CLINICAL TRIAL: NCT05719883
Title: A Prospective, Multi-center, Randomized Controlled Study to Evaluate the Safety and Efficacy of the Maurora® Sirolimus-Eluting Stent Versus the Apollo Stent in Intracranial Atherosclerotic Stenosis(Maurora ICAS Trial)
Brief Title: Evaluating the Safety and Efficacy of the Maurora® DES in ICAS
Acronym: Maurora ICAS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Beijing Tiantan Hospital (Other)
Collaborators: Alain Medical (Beijing) Co., Ltd. (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: QX2022-021-02
Record Dates: First submitted 2023-01-31; First posted 2023-02-09 (Actual); Last update posted 2025-06-26 (Actual); Status verified 2025-06

CONDITIONS: Intracranial Arteriosclerosis; Stroke (CVA) or TIA
Keywords: Intracranial Atherosclerotic stenosis; Drug-eluting stent; Ischemia stroke
MeSH Terms: conditions — Intracranial Arteriosclerosis; Stroke; Ischemic Stroke

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Maurora® Sirolimus Eluting Stent System (Experimental): Device: Maurora® Sirolimus Eluting Stent System A sirolimus eluting intracranial stent system with platform is made of L605 CoCr alloys.
  Interventions: Device: Maurora® Sirolimus Eluting Stent System
- APOLLO™ Intracranial Stent System (Active Comparator): Device: Apollo Intracranial Stent System A 316L stainless steel balloon-expandable intracranial stent system.
  Interventions: Device: APOLLO™ Intracranial Stent System

INTERVENTIONS:
Device: Maurora® Sirolimus Eluting Stent System — The Maurora® for intracranial PTA treatment comprises of a balloon expandable sirolimus eluting stent and a delivery catheter that features a rapid exchange catheter design with a semi-compliant balloon located at its distal end.
  Other Names: Maurora
  Arms: Maurora® Sirolimus Eluting Stent System
Device: APOLLO™ Intracranial Stent System — The Apollo stent system comprises of a balloon expandable stent and a delivery catheter that features a rapid exchange catheter design with a semi-compliant balloon located at its distal end.
  Other Names: APOLLO
  Arms: APOLLO™ Intracranial Stent System

SUMMARY:
The purpose of the RCT trial is to evaluate whether implantation of drug-eluting stent (DES) is more efficacious than bare metal stent (BMS) in prevention of in-stent restenosis (ISR) and improvement of outcomes for symptomatic intracranial atherosclerotic stenosis. This trial is prospective, multi-center, randomized 1:1 single blind trial using Maurora sirolimus eluting stent versus Apollo bare metal stent conducted in approximately 10 interventional neurology centers in China. The study is sponsored by Alain Medical (Beijing) Co., Ltd.

DETAILED DESCRIPTION:
This trial is a prospective, multi-center, 1:1 randomized using drug-eluting (Sirolimus) stent versus bare metal stent (BMS) to treat intracranial stenosis of 70-99% degree. The primary endpoint is in-stent restenosis rate(ISR) within 12 months after revascularization procedure of the qualifying lesion during follow-up.

ELIGIBILITY:
Inclusion Criteria:

1. Age from 18 to 80 years;
2. Symptomatic intracranial atherosclerosis (Definition: Stroke or transient ischemic attack [TIA] associated with intracranial atherosclerosis within 90 days of enrollment);
3. A major intracranial artery (carotid artery, MCA stem [M1], vertebral artery, or basilar artery) with 70% to 99% stenosis on the angiography (According to WASID method);
4. The target lesion length ≤15 mm and the vessel diameter between 2.5mm and 5.0mm, distal vessel diameter >1.5mm;
5. Only one stent planned for the target lesion;
6. A Modified Rankin Score of ≤ 3;
7. Patients understand the purpose and requirements of the study, and can make him/herself understood, and has provided informed consent.

Exclusion Criteria:

1. Ischemic stroke within 2 weeks before the procedure;
2. Tandem extracranial or intracranial stenosis (70%-99%) of the target lesion;
3. Patients with stroke caused by perforating artery occlusion;
4. Severe calcification at target lesion;
5. Any history of brain parenchymal or other intracranial subarachnoid, subdural or extradural hemorrhage in the past 6 weeks;
6. History of stenting or angioplasty of an intracranial artery;
7. Intracranial tumor, aneurysm or intracranial arteriovenous malformation;
8. Intracranial artery stenosis caused by non-atherosclerotic lesions, including: moya-moya disease, vasculitis disease, herpes zoster, varicella-zoster or other viral vascular diseases, neurosyphilis, any other intracranial infections, radiation-induced vascular disease, fibromuscular dysplasia, sickle cell disease, neurofibromatosis, central nervous system benign vascular disease, post-partum vascular disease, suspected vasospasm, suspicious embolism recanalization;
9. Presence of any unequivocal cardiac source of embolism (e.g. atrial fibrillation);
10. Those who cannot tolerate general anesthesia due to insufficiency of cardiac or pulmonary function, not suitable for procedure;
11. Known allergy or contraindication to heparin, aspirin, ticlopidine, ticagrelor, sirolimus, anaesthetics and contrast agents;
12. Severe renal and hepatic insufficiency (ALTor AST > 3x upper limit, creatinine > 1.5x upper limit);
13. Major surgery within the past 30 days or planned within 90 days, or requiring simultaneous intervention to renal artery, iliac artery, and coronary artery;
14. Life expectancy <12 months;
15. Pregnant or lactating women, or planning for pregnancy;
16. Participated in another investigational device or drug study within 30 days;
17. According to the judgement of the investigator, other situations that are not suitable for enrollment.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 156 (Actual)
Dates: Start 2023-02-20 (Actual); Primary Completion 2025-04-30 (Actual); Study Completion 2025-05-15 (Actual)

PRIMARY OUTCOMES:
In-stent restenosis rate(ISR) within 12 months after procedure | 12 months after procedure
  Angiographic evidence of in-stent stenosis ≥50% at 12 months after procedure

SECONDARY OUTCOMES:
Implantation success rate | During the procedure
  Implantation success was defined as successful arrival of stent to the lesion and subsequent release of the stent delivery system.
Technical success rate | During the procedure
  Technical success was defined as successful arrival of stent to the lesion and subsequent release of the stent delivery system with a residual stenosis of <30%.
Clinical success rate | 12 months after procedure
  Clinical success was defined as successful arrival of stent to the lesion and subsequent release of the stent delivery system with a residual stenosis of <30%, and free from major adverse event within 12 months after procedure.
  system with a residual stenosis of <30%
Stroke or death within 30 days after procedure | within 30 days after procedure
  Any stroke included ischemic stroke or/and symptomatic brain hemorrhage and all-cause death.
Stroke in the target vessel territory or death within 30 days after procedure | within 30 days after procedure
  Death or any stroke events related to target vessel after revascularization.
Ischemic stroke in the target vessel territory between 31 day to 1 year after procedure | between 31 day to 1 year after procedure
  Any ischemic stroke events related to target vessel after revascularization.
Ischemic stroke in other vessel territory between 31 day to 1 year after procedure | between 31 day to 1 year after procedure
  Any ischemic stroke events unrelated to target vessel after revascularization.Ischemic stroke is defined as a new focal neurological deficit of sudden onset, that is associated with infarction lesion on CT or MRI. Ischemic strokes are classified as in or out of the territory of the symptomatic intracranial artery.
Any ischemic stroke between 31 day to 1 year after procedure | between 31 day to 1 year after procedure
  Ischemic stroke is defined as a new focal neurological deficit of sudden onset, that is associated with infarction lesion on CT or MRI. Ischemic strokes are classified as in or out of the territory of the symptomatic intracranial artery.
Any subdural, epidural hemorrhage or a systemic hemorrhage between 31 day to 1 year after procedure | between 31 day to 1 year after procedure
  Any subdural or epidural hemorrhage or a systemic hemorrhage is required hospitalization, blood transfusion, or surgery.
Death between 31 day to 1 year after procedure | between 31 day to 1 year after procedure
  All-cause death.
Transient Ischemic Attack within 1 year after the procedure | 1 year after the procedure
  A transient ischemic attack (TIA) is a temporary period of symptoms similar to those of a stroke. A TIA usually lasts only a few minutes up to 24 hours and doesn't cause permanent damage.
Functional outcome measured by the modified Rankin Scale | 1 and 12 months after procedure
  Focus on difference between 1 month and 12 months after procedure. The range of modified Rankin Scale was from 0 to 6. 0-No symptoms; 1-No significant disability; 2-Slight disability; 3-Moderate disability; 4-Moderately severe disability; 5-Severe disability; 6 -Dead. A higher score indicates worse a outcome.

OTHER OUTCOMES:
Complications of stent implantation procedure | 12 months after procedure
  Any complications including vascular complications of assess the intracranial arteries, Allergic reactions or hypersensitivity to agents or device in procedure, complications of intracranial arteries, infection, fever, bleeding and other events.
Stroke | 12 months after procedure
adverse events (AE) and serious adverse events (SAE) | 12 months after procedure

CONTACTS AND LOCATIONS:
Overall Officials: Ning Ma, MD, Principal Investigator — Beijing Tiantan Hospital
Locations (1):
- Beijing Tiantan Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Zhou M, Wang H, Zeng X, Yin P, Zhu J, Chen W, Li X, Wang L, Wang L, Liu Y, Liu J, Zhang M, Qi J, Yu S, Afshin A, Gakidou E, Glenn S, Krish VS, Miller-Petrie MK, Mountjoy-Venning WC, Mullany EC, Redford SB, Liu H, Naghavi M, Hay SI, Wang L, Murray CJL, Liang X. Mortality, morbidity, and risk factors in China and its provinces, 1990-2017: a systematic analysis for the Global Burden of Disease Study 2017. Lancet. 2019 Sep 28;394(10204):1145-1158. doi: 10.1016/S0140-6736(19)30427-1. Epub 2019 Jun 24. PMID 31248666
- [Background] GBD 2016 Stroke Collaborators. Global, regional, and national burden of stroke, 1990-2016: a systematic analysis for the Global Burden of Disease Study 2016. Lancet Neurol. 2019 May;18(5):439-458. doi: 10.1016/S1474-4422(19)30034-1. Epub 2019 Mar 11. PMID 30871944
- [Background] Chimowitz MI, Lynn MJ, Howlett-Smith H, Stern BJ, Hertzberg VS, Frankel MR, Levine SR, Chaturvedi S, Kasner SE, Benesch CG, Sila CA, Jovin TG, Romano JG; Warfarin-Aspirin Symptomatic Intracranial Disease Trial Investigators. Comparison of warfarin and aspirin for symptomatic intracranial arterial stenosis. N Engl J Med. 2005 Mar 31;352(13):1305-16. doi: 10.1056/NEJMoa043033. PMID 15800226
- [Background] Chimowitz MI, Lynn MJ, Derdeyn CP, Turan TN, Fiorella D, Lane BF, Janis LS, Lutsep HL, Barnwell SL, Waters MF, Hoh BL, Hourihane JM, Levy EI, Alexandrov AV, Harrigan MR, Chiu D, Klucznik RP, Clark JM, McDougall CG, Johnson MD, Pride GL Jr, Torbey MT, Zaidat OO, Rumboldt Z, Cloft HJ; SAMMPRIS Trial Investigators. Stenting versus aggressive medical therapy for intracranial arterial stenosis. N Engl J Med. 2011 Sep 15;365(11):993-1003. doi: 10.1056/NEJMoa1105335. Epub 2011 Sep 7. PMID 21899409
- [Background] Shin YS, Kim BM, Suh SH, Jeon P, Kim DJ, Kim DI, Kim BS, Kim KH, Heo JH, Nam HS, Kim YD. Wingspan stenting for intracranial atherosclerotic stenosis: clinical outcomes and risk factors for in-stent restenosis. Neurosurgery. 2013 Apr;72(4):596-604; discussion 604. doi: 10.1227/NEU.0b013e3182846e09. PMID 23277374
- [Background] Jin M, Fu X, Wei Y, Du B, Xu XT, Jiang WJ. Higher risk of recurrent ischemic events in patients with intracranial in-stent restenosis. Stroke. 2013 Nov;44(11):2990-4. doi: 10.1161/STROKEAHA.113.001824. Epub 2013 Aug 20. PMID 23963335